CLINICAL TRIAL: NCT03713541
Title: Identification of Beneficial and Inhibitory Factors for Treatment in Patients With Anorexia Nervosa: A Pathway to Effective Secondary Prevention and Prognostic Improvement
Brief Title: Facilitators and Barriers in Anorexia Nervosa - Treatment Initiation
Acronym: FABIANA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Prof. Dr. Antje Gumz, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: LO 766/16-1m; GU 156
Record Dates: First submitted 2018-08-23; First posted 2018-10-19 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anorexia Nervosa; Feeding and Eating Disorders of Childhood
Keywords: Anorexia nervosa [MeSH]; Feeding and Eating Disorders [MeSH]; women; youth; adolescent; duration of untreated illness (DUI); time-to-treatment [MeSH]; facilitators; barriers; factors; treatment; first treatment initiation
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Anorexia nervosa (AN): Female patients with Anorexia nervosa (AN, ICD-10: F50.0/1) of 14 years and older, receiving an initial treatment due to their AN (start of initial treatment no longer than 3 months ago, inpatient care: at least 7 days inpatient; outpatient care: at least 5 sessions with the same therapist) with sufficient language skills and no serious organic or psychiatric illnesses and no acute suicidality will be consecutively included in the study. No intervention.
  Interventions: Other: No intervention
- Carers of patients with AN: Significant caregivers in AN patients aged 14 to 15 years: parents; in AN patients aged 16 years and over: parents or other significant carer. No intervention.
  Interventions: Other: No intervention
- Physicians of patients with AN: Resident general practitioner, pediatrician, internist or gynecologist with at least one medical patient contact within the last 12 months. No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Survey during normal supply.

SUMMARY:
Anorexia nervosa (AN) is a comparably low-prevalent illness. Chronic courses are often and the mortality rate of patients with AN is higher than in any other mental illness. A major influence on the course of the illness is the interval between the onset of AN symptoms and the beginning of an adequate treatment (duration of untreated illness, DUI). Patients with AN have a better prognosis if treated early. Previous large-scale interventions have not shown the desired positive effects on the DUI. Therefore, an important starting point seems to be a better initial understanding of the factors influencing the DUI, which is the major aim of this project.

The planned mixed-method study is divided in three consecutive sub-studies. The first substudy aims to identify modifiable factors influencing the DUI using semi-structured interviews and a multi-informant approach (patients, carers, physicians). As a result of this qualitative analyses using Grounded Theory the most relevant factors will be determined. The motivation of the second substudy is to condense the factors identified to influence the DUI into a checklist and to conduct a first psychometric evaluation of this newly developed instrument. The third substudy aims to quantitatively determine the magnitude of the effects of a) a priori determined non-modifiable factors and b) the modifiable checklist-factors using a multi-informant approach (planned n for each informant = 130; 13 co-operating specialized clinics and 6 cooperating outpatient partners). Additional outpatient partners may be recruited during the course of the study.

In conclusion, the study aims to derive recommendations for effective secondary prevention. Thereby, the study might ultimately contribute to earlier treatment initiation of patients with AN, and to the prevention of chronic courses and the associated high health care costs and individual burden.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a comparably low-prevalent, yet due to its somatic and mental consequences serious illness. Chronic courses are often and the mortality rate of patients with AN is higher than in any other mental illness.

A major influence on the course of the illness is the interval between the onset of AN symptoms and the beginning of an adequate treatment (duration of untreated illness, DUI). That is, patients with AN have a better prognosis if treated early. Previous large-scale interventions have not shown the desired positive effects on the DUI. Therefore, an important starting point seems to be a better initial understanding of the factors influencing the DUI, which is the major aim of this project. Based on this evidence, this study aims to derive recommendations for effective secondary prevention.

To our very best knowledge this is the first study investigating factors influencing the DUI using a multi-informant strategy, that is exploring the perspective of patients with AN, their significant carers and involved physicians. Furthermore, the study will avoid the confounding of patients with different eating disorder diagnoses, i.e. it will include exclusively patients with AN. Finally, there will be a clear focus on factors which are modifiable and precise in their definition.

The planned mixed-method study is divided in three consecutive sub-studies. The first substudy aims to identify modifiable factors influencing the DUI using semi-structured interviews and a multi-informant approach (patients, carers, physicians). As a result of this qualitative analyses using Grounded Theory the most relevant factors will be determined. The motivation of the second substudy is to condense the factors identified to influence the DUI into a checklist and to conduct a first psychometric evaluation of this newly developed instrument. The third substudy aims to quantitatively determine the magnitude of the effects of a) a priori determined non-modifiable factors and b) the modifiable checklist-factors using a multi-informant approach (planned n for each informant = 130; 13 co-operating specialized clinics and 6 cooperating outpatient partners). Additional outpatient partners may be recruited during the course of the study.

In conclusion, the study aims to derive recommendations for effective secondary prevention. Thereby, the study might ultimately contribute to earlier treatment initiation of patients with AN, and to the prevention of chronic courses and the associated high health care costs and individual burden.

ELIGIBILITY:
AN patients

Inclusion criteria

* Female patients, 14 years and older
* Treatment diagnosis anorexia nervosa (ICD-10: F50.0/1)
* Initial treatment (start of initial treatment no longer than 3 months ago)
* Inpatient care: at least 7 days inpatient
* Outpatient care: at least 5 sessions with the same therapist

Exclusion criteria

* Insufficient language skills
* Serious organic or psychiatric illnesses
* Acute suicidality

Significant caregiver

Inclusion criteria

* in AN patients aged 14 to 15 years: parents ; in AN patients aged 16 years and over: parents or other significant carer
* Informed consent
* Consent of the patient

Exclusion criteria - Insufficient language skills

Physician

Inclusion criteria

* Resident general practitioner, pediatrician, internist or gynecologist
* At least one medical patient contact within the last 12 months
* Informed consent
* Consent of the patient and release from confidentiality

Exclusion criteria

- Insufficient language skills

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AN will be recruited from n=13 inpatient clinics with special treatment units/specialized inpatient units and n=6 outpatient psychotherapists specialized for eating disorders.
  Additional outpatient partner may be recruited during the course of the study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Duration of untreated illness (DUI in months) | from date of study enrolment up to 12 weeks
  DUI (defined as the time between occurence of first symptoms and treatment) is assessed retrospectively and cross-sectional using standardized interviews and paper-and-pencil questionnaires.

SECONDARY OUTCOMES:
Duration of first contact (DUC in month) | from date of study enrolment up to 12 weeks
  DUC is assessed cross-sectional (retrospectively) using standardized interviews and paper-and-pencil questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Gumz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Bernd Loewe, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (18):
- Germany (18):
  - Schön Clinic Roseneck, Prien am Chiemsee, Bavaria
  - Schön Clinic Bad Bramstedt, Bad Bramstedt, Schleswig-Holstein
  - Curtius-Clinic, Specialist Clinic for Psychosomatics and Psychotherapeutic Medicine, Malente, Schleswig-Holstein
  - Schön Clinic Bad Arolsen, Bad Arolsen
  - Clinic Lüneburger Heide, Bad Bevensen
  - MediClin Seepark Clinic, Bodenteich
  - Timmermann & Partner, Medical care center for physical and mental health, Cuxhaven
  - Department of Child and Adolescent Psychiatry of the University Medical Center Hamburg-Eppendorf (UKE), Hamburg
  - Local psychotherapists, Hamburg
  - Behavior therapy Falkenried MVZ GmbH, Hamburg
  - VT Falkenried Training and Education, Hamburg
  - Department of Psychosomatic Medicine and Psychotherapy, Asklepios West Clinic Hamburg, Hamburg
  - Schön Clinic Eilbek, Hamburg
  - Schön Clinic Hamburg Eilbek, Hamburg
  - Institute for Behavior Therapy Education Hamburg (IVAH), Hamburg
  - Asklepios Clinic Nord - Ochsenzoll, Hamburg
  - University Clinic Regensburg, Regensburg
  - Evangelic hospital Ginsterhof HmbH, Rosengarten

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reuter L, Kastner D, Schmidt J, Weigel A, Voderholzer U, Seidel M, Schwennen B, Fehrs H, Lowe B, Gumz A. The development and psychometric evaluation of FABIANA-checklist: a scale to assess factors influencing treatment initiation in anorexia nervosa. J Eat Disord. 2021 Nov 3;9(1):144. doi: 10.1186/s40337-021-00490-w. PMID 34732246
- [Derived] Kastner D, Weigel A, Buchholz I, Voderholzer U, Lowe B, Gumz A. Facilitators and barriers in anorexia nervosa treatment initiation: a qualitative study on the perspectives of patients, carers and professionals. J Eat Disord. 2021 Feb 27;9(1):28. doi: 10.1186/s40337-021-00381-0. PMID 33640028
- [Derived] Kastner D, Buchholz I, Weigel A, Brunner R, Voderholzer U, Gumz A, Lowe B. Facilitators and barriers in anorexia nervosa treatment initiation (FABIANA): study protocol for a mixed-methods and multicentre study. BJPsych Open. 2019 Oct 21;5(6):e92. doi: 10.1192/bjo.2019.77. PMID 31631825